CLINICAL TRIAL: NCT06402032
Title: Clinical and Histological Evaluation of Hesperidin Versus Mineral Trioxide Aggregate (MTA) as a Direct Pulp Capping Material: A Randomized Controlled Trial
Brief Title: Clinical and Histological Evaluation of Hesperidin as a Direct Pulp Capping Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Kamal Eldin, Lecturer, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hesperidin_MTA
Record Dates: First submitted 2024-04-30; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pulp Exposure, Dental; Dental Pulp Capping
MeSH Terms: conditions — Dental Pulp Exposure | interventions — Hesperidin; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hesperidin (Experimental)
  Interventions: Other: Hesperidin
- Mineral trioxide aggregate (MTA) (Active Comparator)
  Interventions: Other: Mineral Trioxide Aggregate (MTA)

INTERVENTIONS:
Other: Hesperidin — Hesperidin is a natural flavonoid with well-known of its anti-inflammatory properties in many disease. Hesperidin in previous studies has been documented to reduce inflammation as well as pain through suppression of cytokine production, NF-κB activity, and oxidative stress. Hesperidin, as a natural product, have been considered as a promising pulp capping material in several invitro and animal studies. However, the regenerative effect of hesperidin as pulp capping material in human teeth has not yet been reported.
  Arms: Hesperidin
Other: Mineral Trioxide Aggregate (MTA) — Mineral trioxide aggregate is a cementitious material having various advantages as it is biocompatible, bioactive, osteo-inductive, non-resorbable material with exciting clinical applications, stimulating reparative continuous dentin formation along with maintaining the integrity of the pulp. Moreover, mineral trioxide aggregate provides seal to tooth structure and is of high strength. It is considered the gold standard material for direct pulp capping.
  Arms: Mineral trioxide aggregate (MTA)

SUMMARY:
Direct pulp capping technique is one of the oldest known treatments for exposed pulp tissue, and there is a continuous requirement for the most efficient materials to be used in this approach. Successful pulp capping is the usual way to preserve the vitality of tooth and avoid root canal treatment or surgical tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene,
* Sound wisdom teeth with closed apices with normal pulp vitality response
* No periodontal disease or periapical lesions on periapical radiograph
* Cooperative patients approving to participate in the study

Exclusion Criteria:

* Medically compromised participants
* Evidence of parafunctional habits
* Heavy smokers
* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis
* Severe periodontal problems or pathological periapical changes
* Teeth with open apex or pulp calcification

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Success Rate (Clinical evaluation) | after 12 weeks
  Teeth with vital pulp (numerical values with electric pulp tester) and absence of clinical signs/symptoms (Visual Analog Score for pain) as one reported value indicating clinical success rate (%)

SECONDARY OUTCOMES:
Histomorphometric analysis (Histologic evaluation) | after 12 weeks
  Thickness of formed dentin bridge (μm)
Histomorphometric analysis (Histologic evaluation) | after 12 weeks
  Number of inflammatory cells in pulp (scores for Inflammation intensity/extensity)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt